CLINICAL TRIAL: NCT02021656
Title: A Phase 3b, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Ledipasvir Fixed-Dose Combination in Treatment-Naïve and Treatment-Experienced Subjects With Chronic Genotype 1 HCV Infection
Brief Title: Efficacy and Safety of Ledipasvir/Sofosbuvir Fixed-Dose Combination in Participants With Chronic Genotype 1 HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-0131
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2019-01

CONDITIONS: Chronic HCV Infection
MeSH Terms: interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- LDV/SOF (Experimental): Treatment-experienced and treatment-naive participants will receive LDV/SOF for 12 weeks.
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily without regard to food
  Other Names: Harvoni®; GS-5885/GS-7977

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of treatment with ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) in treatment-naive and treatment-experienced participants with chronic genotype 1 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV RNA ≥ 10^4 IU/mL at screening
* HCV treatment-naive, as defined as no prior exposure to any interferon (IFN) or other approved or experimental HCV-specific direct-acting antiviral agent; OR HCV treatment-experienced with medical records that include sufficient detail of prior IFN-based treatment to allow for categorization of prior response as either intolerant, non-responder, or experienced viral breakthrough or relapse.
* Genotype 1 HCV at screening
* HCV infection documented by anti-HCV antibody test, genotyping test, or liver biopsy

Key Exclusion Criteria:

* Pregnant or nursing female
* Chronic liver disease of a non-HCV etiology
* Current or prior history of any clinically-significant illness (other than HCV)
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2013-12-10 (Actual); Primary Completion 2017-07-08 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (26):
- China (12):
  - Beijing
  - Chongqing
  - Guangdong
  - Guangxi
  - Hubei
  - Hunan
  - Jiangxi
  - Jilin
  - Shandong
  - Shanghai
  - Shijiazhuang
  - Sichuan
- South Korea (7):
  - Ansan-si, Gyeonggi-do
  - Bucheon-si, Gyeonggi-do
  - Incheon, Gyeonggi-do
  - Seongnam-si, Gyeonggi-do
  - Busan
  - Daegu
  - Seoul
- Taiwan (7):
  - Changhua
  - Kaohsiung City
  - Keelung
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Wei L, Xie Q, Hou JL, et al. Safety and Efficacy of Ledipasvir/Sofosbuvir in a Genotype 1 HCV Infected Chinese Population: Results from a Phase 3 Clinical Trial. Poster No. 1191, AASLD 2017.
- [Result] Lim YS, Ahn SH, Lee KS, Paik SW, Lee YJ, Jeong SH, Kim JH, Yoon SK, Yim HJ, Tak WY, Han SY, Yang JC, Mo H, Garrison KL, Gao B, Knox SJ, Pang PS, Kim YJ, Byun KS, Kim YS, Heo J, Han KH. A phase IIIb study of ledipasvir/sofosbuvir fixed-dose combination tablet in treatment-naive and treatment-experienced Korean patients chronically infected with genotype 1 hepatitis C virus. Hepatol Int. 2016 Nov;10(6):947-955. doi: 10.1007/s12072-016-9726-5. Epub 2016 May 20. PMID 27198664
- [Result] Chuang WL, Chien RN, Peng CY, Chang TT, Lo GH, Sheen IS, Wang HY, Chen JJ, Yang JC, Knox SJ, Gao B, Garrison KL, Mo H, Pang PS, Hsu YC, Hu TH, Chu CJ, Kao JH. Ledipasvir/sofosbuvir fixed-dose combination tablet in Taiwanese patients with chronic genotype 1 hepatitis C virus. J Gastroenterol Hepatol. 2016 Jul;31(7):1323-9. doi: 10.1111/jgh.13305. PMID 26841930
- [Result] Wei L, Xie Q, Hou JL, et al. Safety and Efficacy of Ledipasvir/Sofosbuvir in a Genotype 1 HCV Infected Chinese Population: Results from a Phase 3 Clinical Trial., [Abstract 1191]. The Liver Meeting® 2017 - The 68th Annual Meeting of the American Association for the Study of Liver Diseases (AASLD); 2017 20-24 October; Washington, D. C.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Mainland China (referred to as China throughout this results record), Korea, and Taiwan. The first participant was screened on 10 December 2013. The last study visit occurred on 29 September 2017.
Pre-assignment Details: 416 participants were screened.
Groups:
- LDV/SOF (Overall): Ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet once daily administered without regard to food for 12 weeks in treatment-experienced and treatment-naive participants in China, Korea, and Taiwan
Period: Overall Study
Arm/Group | LDV/SOF (Overall)
Started | 384
Completed | 378
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrew Consent | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study
Groups:
- LDV/SOF: LDV/SOF (90/400 mg) FDC tablet administered once daily without regard to food for 12 weeks in treatment-experienced and treatment-naive participants in China, Korea, and Taiwan
Arm/Group | LDV/SOF
Number analyzed (Participants) | 384
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202
  Male | 182
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race Subcategory: Chinese | 207
  Race Subcategory: Korean | 93
  Race Subcategory: Taiwanese | 83
  Race Subcategory: Other (Taiwanese- Chinese) | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 384
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 93
  China | 206
  Taiwan | 85
IL28B [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 286
    CT | 95
    TT | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, < 25 IU/mL in Korea and Taiwan and < 15 IU/mL in China) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full analysis set: participants who were enrolled and received at least 1 dose of study drug, and have chronic genotype 1 HCV infection.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- LDV/SOF: China: LDV/SOF (90/400 mg) FDC tablet administered once daily in treatment-experienced and treatment-naive participants in China without regard to food for 12 weeks
- LDV/SOF: Overall: LDV/SOF (90/400 mg) FDC tablet administered once daily in treatment-experienced and treatment-naive participants in China, Korea, and Taiwan without regard to food for 12 weeks
Arm/Group | LDV/SOF: China | LDV/SOF: Overall
Number analyzed (Participants) | 206 | 384
Percentage of participants | 100.0 [98.2 to 100.0] | 99.2 [97.7 to 99.8]
Statistical Analysis 1: Comparison: LDV/SOF: China; A sample size of 100 Chinese participants in the treatment naive group provided at least 90% power to detect a 17% improvement in SVR12 rate from the historical control rate of 57% using 2-sided exact one-sample binomial test at significant level of 0.05; Test type: Superiority; p < 0.001, Binomial Exact Test

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF: China | LDV/SOF: Overall
Number analyzed (Participants) | 206 | 384
percentage of participants | 0 | 0.5

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- LDF/SOF: Overall: LDV/SOF (90/400 mg) FDC tablet administered once daily in treatment-experienced and treatment-naive participants in Korea and Taiwan without regard to food for 12 weeks.
Arm/Group | LDV/SOF: China | LDF/SOF: Overall
Number analyzed (Participants) | 206 | 384
percentage of participants
  SVR4 | 100.0 [98.2 to 100.0] | 99.2 [97.7 to 99.8]
  SVR24 | 100.0 [98.2 to 100.0] | 99.0 [97.4 to 99.7]

4. Secondary Outcome: Percentage of Participants Experiencing Viral Breakthrough
Description: Viral breakthrough were defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) during treatment, but did not achieve a sustained virologic response (SVR).
Time Frame: Up to 12 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- LDF/SOF: Overall: LDV/SOF (90/400 mg) FDC tablet administered once daily in treatment-experienced and treatment-naive participants in China, Korea, and Taiwan without regard to food for 12 weeks.
Arm/Group | LDV/SOF: China | LDF/SOF: Overall
Number analyzed (Participants) | 206 | 384
percentage of participants | 0 | 0

5. Secondary Outcome: Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse is defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) within 4 weeks of end of treatment, but did not achieve an SVR.
Time Frame: Week 12 to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF: China | LDF/SOF: Overall
Number analyzed (Participants) | 206 | 384
percentage of participants | 0 | 0.5

6. Secondary Outcome: HCV RNA and Change From Baseline in HCV RNA Through Week 12 for China Only
Time Frame: Baseline; Week 12
Population: Only Chinese participants in the Full Analysis set were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF: China
Number analyzed (Participants) | 206
log10 IU/mL
  Baseline | 6.31 (0.633)
  Change at Week 12 | -5.16 (0.633)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study
Groups:
- LDV/SOF (Overall): LDV/SOF (90/400 mg) FDC tablet administered once daily without regard to food for 12 weeks in treatment-experienced and treatment-naive participants in China, Korea, and Taiwan
Arm/Group | LDV/SOF (Overall)
All-Cause Mortality (participants affected / at risk) | 0/384
Serious Adverse Events (participants affected / at risk) | 7/384
Other Adverse Events (participants affected / at risk) | 105/384
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (Overall) (N=384)
Erysipelas (Infections and infestations) | 1
Bone contusion (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adenomyosis (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (Overall) (N=384)
Upper respiratory tract infection (Infections and infestations) | 42
Viral upper respiratory tract infection (Infections and infestations) | 44
Headache (Nervous system disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Original (2013-05-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT02021656/Prot_000.pdf
  • Study Protocol: Amendment 2 (2014-08-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT02021656/Prot_001.pdf
  • Study Protocol: Amendment 3 (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT02021656/Prot_002.pdf
  • Statistical Analysis Plan (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT02021656/SAP_003.pdf